CLINICAL TRIAL: NCT04457908
Title: the Effectiveness and Cost Effectiveness in Screening Gait Disorder of Silent Cerebrovascular Disease Assisted by Artificial Intelligent System and Clinical Doctors - A Randomized Parallel-controlled Study
Brief Title: The Effectiveness and Cost Effectiveness of Intelligent Assessment of Gait Disorder in Silent Cerebrovascular Disease
Acronym: ACCURATE-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fudan University (Other); The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2018YFC1312900-05
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2019-10

CONDITIONS: Silent Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intelligent (Other): receive the neurological function assessment by artificial intelligence
  Interventions: Diagnostic Test: intelligent assessment
- manual (No Intervention): receive the neurological function assessment by doctor

INTERVENTIONS:
Diagnostic Test: intelligent assessment — intelligent neurological function assessment
  Arms: intelligent

SUMMARY:
This is a multi-center, randomized, double-blind, parallel-controlled, prospective study to compare the effectiveness and cost-effectiveness of intelligent and doctor groups for gait disorder screening.

Clinical data, including demographic characteristics, socioeconomic level, medical history, assessment of neurological function, laboratory tests, imaging tests, health service utilization, and costs will be collected from the subjects. All subjects will be divided into an intelligent group and a doctor group according to a 1:1 ratio. The intelligent group will undergo intelligent system evaluation, and the doctor group will undergo the clinician's conventional treatment process. At the same time, all the subjects will undergo gold-standard panel gait and cognitive rating scale assessments.

DETAILED DESCRIPTION:
All subjects in the intelligent group will undergo tests to evaluate their nervous system function, including the timed up-and-go test, mini-cognitive assessment, and sentence repetition. Subjects will be recorded using a camera and microphone. The intelligent system uses the built-in intelligent algorithm to analyze the gait video, sound, and picture to provide information on gait features (stand-up time, turnaround time, stride length, step velocity, stride length, step width, etc.), language features (pronunciation, intonation, word order, language accuracy, language fluency, etc.), and clock features (contour, numbers, pointers, etc.).

All subjects in the doctor group will consult with a doctor in the non-intelligent group according to the routine treatment procedure. Doctors in the non-intelligent group are required to be internal medicine clinicians with intermediate title or below, and they should have registered their qualifications, relevant knowledge and training experience, educational background, and other information in the early stage of the study. The doctors in the non-intelligent group will make clinical diagnoses for the subjects based on routine medical operations such as a history of the present illness, previous history, and physical examination, and the data in medical records in the outpatient department will help determine whether the subjects have gait disorders.

All subjects' walking videos will be assessed by the gold-standard panel, which will consist of 2 experts of movement disorders. If there is any difference, a third expert will be included in the evaluation. According to the clinical experience, the expert doctors will evaluate the subjects' gait, and the results will be divided into normal gait and abnormal gait.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 60 and 85 years.
2. Diagnosed with silent cerebrovascular disease/silent stroke, which is consistent with the 2016 statement issued by the American Heart Association (AHA) and American Stroke Association (ASA):

   1. No previous clear history of stroke and no clinical symptoms or mild clinical symptoms that fail to attract clinical attention;
   2. Cranial MRI showing at least one of the following within 5 years: lacunar infarct of vascular origin, white matter hyperintensity of vascular origin, cerebral microbleeds;
3. Consciousness and ability to complete cognitive assessment
4. Ability to stand and walk independently and complete gait assessment without assistance from others.
5. Ability to sign the informed consent.

Exclusion Criteria:

1. Intracranial lesions that have been clearly diagnosed as demyelination disease, white matter dystrophy, intracranial space-occupying lesions, or autoimmune encephalitis.
2. Gait disorder that has been diagnosed as Parkinson's disease, normal cranial hydrocephalus, an otogenic disease, subacute combined degeneration, peripheral neuropathy, osteoarthritis, or lumbar disease.
3. Cognitive disorders that have been diagnosed, such as Alzheimer's disease, frontotemporal dementia, Lewy body dementia, etc.
4. Severe neurological diseases such as previous cerebral trauma, epilepsy, and myelopathy, etc.
5. Severe cardiovascular complications and intolerance to the assessment
6. Severe visual or hearing impairment, aphasia, cognitive disorder, gait disorder, etc., that results in the inability to cooperate for cognitive and gait assessment
7. Refusal to participate in the study
8. Other anomalies that could not be included in the exclusion criteria, but are considered inappropriate to be included in this study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | baseline
  Compared with the gold standard panel of neurology, the sensitivity of the intelligent system and clinicians to screen for gait disorders

SECONDARY OUTCOMES:
Specificity | baseline
  the specificity of the intelligent system and clinicians to screen for gait disorders
Coincidence | baseline
  the coincidence of the intelligent system and clinicians to screen for gait disorders
Yoden index | baseline
  the Yoden index of the intelligent system and clinicians to screen for gait disorders
Positive predictive value and negative predictive value | baseline
  the positive predictive value and negative predictive value of the intelligent system and clinicians at different levels to screen for gait disorders
Cost and cost-effectiveness | baseline
  Health care utilization and costs will be collected to calculate direct and indirect costs of the intelligent system and clinicians to screen for gait disorders, and the incremental cost-effectiveness ratio (ICER) will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ding, MD, Study Director — Shanghai Zhongshan Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poels MM, Steyerberg EW, Wieberdink RG, Hofman A, Koudstaal PJ, Ikram MA, Breteler MM. Assessment of cerebral small vessel disease predicts individual stroke risk. J Neurol Neurosurg Psychiatry. 2012 Dec;83(12):1174-9. doi: 10.1136/jnnp-2012-302381. Epub 2012 Aug 23. PMID 22917672
- [Background] Kim BJ, Lee SH. Prognostic Impact of Cerebral Small Vessel Disease on Stroke Outcome. J Stroke. 2015 May;17(2):101-10. doi: 10.5853/jos.2015.17.2.101. Epub 2015 May 29. PMID 26060797
- [Background] Sachdev PS, Wen W, Christensen H, Jorm AF. White matter hyperintensities are related to physical disability and poor motor function. J Neurol Neurosurg Psychiatry. 2005 Mar;76(3):362-7. doi: 10.1136/jnnp.2004.042945. PMID 15716527
- [Background] Murray ME, Senjem ML, Petersen RC, Hollman JH, Preboske GM, Weigand SD, Knopman DS, Ferman TJ, Dickson DW, Jack CR Jr. Functional impact of white matter hyperintensities in cognitively normal elderly subjects. Arch Neurol. 2010 Nov;67(11):1379-85. doi: 10.1001/archneurol.2010.280. PMID 21060015
- [Background] Wakefield DB, Moscufo N, Guttmann CR, Kuchel GA, Kaplan RF, Pearlson G, Wolfson L. White matter hyperintensities predict functional decline in voiding, mobility, and cognition in older adults. J Am Geriatr Soc. 2010 Feb;58(2):275-81. doi: 10.1111/j.1532-5415.2009.02699.x. Epub 2010 Jan 26. PMID 20374403
- [Background] Debette S, Markus HS. The clinical importance of white matter hyperintensities on brain magnetic resonance imaging: systematic review and meta-analysis. BMJ. 2010 Jul 26;341:c3666. doi: 10.1136/bmj.c3666. PMID 20660506
- [Background] Brickman AM, Provenzano FA, Muraskin J, Manly JJ, Blum S, Apa Z, Stern Y, Brown TR, Luchsinger JA, Mayeux R. Regional white matter hyperintensity volume, not hippocampal atrophy, predicts incident Alzheimer disease in the community. Arch Neurol. 2012 Dec;69(12):1621-7. doi: 10.1001/archneurol.2012.1527. PMID 22945686
- [Background] Maillard P, Carmichael O, Fletcher E, Reed B, Mungas D, DeCarli C. Coevolution of white matter hyperintensities and cognition in the elderly. Neurology. 2012 Jul 31;79(5):442-8. doi: 10.1212/WNL.0b013e3182617136. Epub 2012 Jul 18. PMID 22815562
- [Background] Smith EE, Saposnik G, Biessels GJ, Doubal FN, Fornage M, Gorelick PB, Greenberg SM, Higashida RT, Kasner SE, Seshadri S; American Heart Association Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Functional Genomics and Translational Biology; and Council on Hypertension. Prevention of Stroke in Patients With Silent Cerebrovascular Disease: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Feb;48(2):e44-e71. doi: 10.1161/STR.0000000000000116. Epub 2016 Dec 15. PMID 27980126
- [Background] Leary MC, Saver JL. Annual incidence of first silent stroke in the United States: a preliminary estimate. Cerebrovasc Dis. 2003;16(3):280-5. doi: 10.1159/000071128. PMID 12865617
- [Background] Kim YJ, Kwon HK, Lee JM, Cho H, Kim HJ, Park HK, Jung NY, San Lee J, Lee J, Jang YK, Kim ST, Lee KH, Choe YS, Kim YJ, Na DL, Seo SW. Gray and white matter changes linking cerebral small vessel disease to gait disturbances. Neurology. 2016 Mar 29;86(13):1199-207. doi: 10.1212/WNL.0000000000002516. Epub 2016 Mar 2. PMID 26935893
- [Background] de Laat KF, van Norden AG, Gons RA, van Oudheusden LJ, van Uden IW, Bloem BR, Zwiers MP, de Leeuw FE. Gait in elderly with cerebral small vessel disease. Stroke. 2010 Aug;41(8):1652-8. doi: 10.1161/STROKEAHA.110.583229. Epub 2010 Jun 24. PMID 20576951
- [Background] Montero-Odasso MM, Sarquis-Adamson Y, Speechley M, Borrie MJ, Hachinski VC, Wells J, Riccio PM, Schapira M, Sejdic E, Camicioli RM, Bartha R, McIlroy WE, Muir-Hunter S. Association of Dual-Task Gait With Incident Dementia in Mild Cognitive Impairment: Results From the Gait and Brain Study. JAMA Neurol. 2017 Jul 1;74(7):857-865. doi: 10.1001/jamaneurol.2017.0643. PMID 28505243
- [Background] Wardlaw JM, Smith EE, Biessels GJ, Cordonnier C, Fazekas F, Frayne R, Lindley RI, O'Brien JT, Barkhof F, Benavente OR, Black SE, Brayne C, Breteler M, Chabriat H, Decarli C, de Leeuw FE, Doubal F, Duering M, Fox NC, Greenberg S, Hachinski V, Kilimann I, Mok V, Oostenbrugge Rv, Pantoni L, Speck O, Stephan BC, Teipel S, Viswanathan A, Werring D, Chen C, Smith C, van Buchem M, Norrving B, Gorelick PB, Dichgans M; STandards for ReportIng Vascular changes on nEuroimaging (STRIVE v1). Neuroimaging standards for research into small vessel disease and its contribution to ageing and neurodegeneration. Lancet Neurol. 2013 Aug;12(8):822-38. doi: 10.1016/S1474-4422(13)70124-8. PMID 23867200
- [Result] Vermeer SE, Longstreth WT Jr, Koudstaal PJ. Silent brain infarcts: a systematic review. Lancet Neurol. 2007 Jul;6(7):611-9. doi: 10.1016/S1474-4422(07)70170-9. PMID 17582361
- [Result] Vermeer SE, Hollander M, van Dijk EJ, Hofman A, Koudstaal PJ, Breteler MM; Rotterdam Scan Study. Silent brain infarcts and white matter lesions increase stroke risk in the general population: the Rotterdam Scan Study. Stroke. 2003 May;34(5):1126-9. doi: 10.1161/01.STR.0000068408.82115.D2. Epub 2003 Apr 10. PMID 12690219
- [Result] Verghese J, Lipton RB, Hall CB, Kuslansky G, Katz MJ, Buschke H. Abnormality of gait as a predictor of non-Alzheimer's dementia. N Engl J Med. 2002 Nov 28;347(22):1761-8. doi: 10.1056/NEJMoa020441. PMID 12456852
- [Result] Dumurgier J, Artaud F, Touraine C, Rouaud O, Tavernier B, Dufouil C, Singh-Manoux A, Tzourio C, Elbaz A. Gait Speed and Decline in Gait Speed as Predictors of Incident Dementia. J Gerontol A Biol Sci Med Sci. 2017 May 1;72(5):655-661. doi: 10.1093/gerona/glw110. PMID 27302701
- [Derived] Fei B, Zhao J, Li X, Tang Y, Qin G, Zhang W, Ding J, Hu M, Wang X. Randomised parallel trial on the effectiveness and cost-effectiveness in screening gait disorder of silent cerebrovascular disease assisted by artificial intelligent system versus clinical doctors (ACCURATE-1): study protocol. BMJ Open. 2022 Mar 24;12(3):e055880. doi: 10.1136/bmjopen-2021-055880. PMID 35332042